CLINICAL TRIAL: NCT00354588
Title: Observational Study on the Prognostic Significance (Renal and Cardiovascular) of Arterial Stiffness and Arterial Wave Reflections in Patients With Mild to Moderate Renal Impairment
Brief Title: Arterial Stiffness, Wave Reflections and Renal Failure
Status: Completed | Type: Observational
Sponsor: Klinikum Wels-Grieskirchen (Other)
Responsible Party: Thomas Weber, MD, Klinikum Wels-Grieskirchen
Other Study IDs: WelsEK 206
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Renal Failure; Arterial Stiffness; Arterial Wave Reflections
Keywords: chronic renal failure; arterial stiffness; arterial wave reflections
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
1. Cardiovascular risk is high in patients with renal failure.
2. Cross-sectional studies have indicated a relationship between arterial stiffness and renal function. However, there are no prospective longitudinal studies in the literature.
3. In dialysis patients, arterial stiffness as well as wave reflections, predict mortality. However, there are no data on patients with mild-to-moderate renal impairment available.
4. Therefore, we designed a study to test the hypothesis that: a) measures of arterial stiffness and wave reflections predict the progression of renal impairment in patients with mild-to-moderate renal failure; and b) measures of arterial stiffness and wave reflections predict cardiovascular events in patients with mild-to-moderate renal failure

ELIGIBILITY:
Inclusion Criteria:

* chronic renal failure patients (KDOQI III, IV) undergoing regular control visits at our nephrology department
* > 19 years
* written informed consent

Exclusion Criteria:

* atrial fibrillation
* valvular heart disease
* severely impaired systolic function
* no informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic renal failure
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2006-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
renal endpoint
  doubling serum creatinine, need for dialysis, renal transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Weber, MD, Principal Investigator — Cardiology Department, Klinikum Wels, Austria; Manfred Wallner, MD, Principal Investigator — Nephrology Department, Klinikum Wels, Austria
Locations (1):
- Cardiology and Nephrology Department Klinikum Wels, Wels, Austria